CLINICAL TRIAL: NCT04679935
Title: A 52-week, Two Arm, Randomized, Open-label, Multicenter Study Assessing the Efficacy and Safety of Two Different Brolucizumab 6 mg Dosing Regimens for Patients With Suboptimal Anatomically Controlled Neovascular Age-related Macular Degeneration
Brief Title: Efficacy and Safety of Two Different Brolucizumab 6 mg Dosing Regimens in Neovascular Age-related Macular Degeneration
Acronym: FALCON
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRTH258ADE01; 2019-004767-53 (EudraCT Number)
Record Dates: First submitted 2020-12-03; First posted 2020-12-22 (Actual); Results first posted 2025-01-27 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Age-related Macular Degeneration
Keywords: neovascular age-related macular degeneration; anti-VEGF; choroidal neovascularization; brolucizumab; loading vs. non-loading; Macular degeneration; age-related macular degeneration (ARMD); vision loss; macula damage; retina damage; dry macular degeneration; wet macular degeneration; Subfoveal choroidal neovascularization (CNV) secondary to age-related macular degeneration; Retinal Degeneration; Retinal Diseases; Eye Diseases
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization; Vision Disorders; Geographic Atrophy; Wet Macular Degeneration; Retinal Degeneration; Retinal Diseases; Eye Diseases | interventions — brolucizumab

STUDY DESIGN:
Intervention Model Description: two arm, multicenter
Masking Description: open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brolucizumab 6 mg non-loading (Experimental): One initial injection followed by treatment every 12 weeks.
  Interventions: Biological: Brolucizumab
- Brolucizumab 6 mg loading (Experimental): 3 x 4-weekly injections followed by treatment every 12 weeks.
  Interventions: Biological: Brolucizumab

INTERVENTIONS:
Biological: Brolucizumab — Intravitreal injection
  Other Names: RTH258, Beovu

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of two different brolucizumab 6 mg dosing regimens in patients with visual impairment due to age-related macular degeneration (AMD) who have previously received anti-VEGF (vascular endothelial growth factor) treatment.

DETAILED DESCRIPTION:
This study was a 52-week randomized, open-label, multi-center, two-arm study for pretreated patients with suboptimal anatomically controlled nAMD. Patients who consented were screened to evaluate eligibility. Eligible patients were randomized in a 1:1 ratio to one of the two treatment arms:

* Brolucizumab 6 mg "loading arm": 1 loading injection every 4 weeks for 3 consecutive injections (baseline, weeks 4 and 8) followed by an injection every 12 weeks.
* Brolucizumab 6 mg "non-loading arm": one initial injection followed by an injection every 12 weeks

There were three periods in this study:

* Screening period: from day -14 to baseline
* Open-label treatment period: from baseline (day 1) to week 48
* Post-treatment follow-up period: from week 48 to week 52

In both study arms, treatment intervals after the initiation phase were either 8 weeks or 12 weeks depending on disease activity status. More frequent injections, i.e., treatment intervals of < 8 weeks were not allowed after the initiation phase.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 50 years of age at screening
* Active choroidal neovascularization (CNV) secondary to AMD that affects the central subfield, including retinal angiomatous proliferation (RAP) with a CNV component, confirmed by presence of active leakage from CNV seen by fluorescein angiography and sequellae of CNV, e.g. pigment epithelial detachment (PED), subretinal or sub-retinal pigment epithelium (sub-RPE) hemorrhage, blocked fluorescence, macular edema (intraretinal fluid (IRF) and/or subretinal fluid (SRF) and/or sub-retinal pigment epithelium (sub-RPE) fluid that affects the central subfield, as seen by spectral domain optical coherence tomography (SD-OCT)) at screening, as confirmed by central reading center (study eye). If active CNV according to the above explained activity criteria is not detectable in screening image data (no IRF and no SRF), presence of residual and/or recurrent fluid (IRF and / or SRF) within the last 6 months before baseline visit is also considered eligible. In this case, historical images must be submitted for analysis by the central reading center.
* Pretreatment with any anti-VEGF drug for a maximum of five years (60 months). Patients should have shown functional and/or anatomical treatment response to the pretreatment(s), prior to participating in this study.
* The treatment initiation phase with the current anti-VEGF must have been completed for at least 6 months with continuous treatment in a ≥ q4w to ≤ q12w injection interval (±2-day window, i.e., 26 to 86 days inclusive) before the baseline visit. At least 4 weeks (minimum 26 days) must have passed between the last anti-VEGF pretreatment and baseline.
* Best-corrected visual acuity (BCVA) score between 83 and 38 letters, inclusive, using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts at both screening and baseline visit (study eye)

Exclusion Criteria:

* Any active intraocular or periocular infection or active intraocular inflammation, at screening or baseline (study eye)
* Uncontrolled glaucoma defined as intraocular pressure (IOP) > 25 mmHg on medication, or according to investigator's judgement, at screening or baseline (study eye)
* Presence of amblyopia, amaurosis or ocular disorders in the fellow eye with BCVA <20/200 at screening (except when due to conditions whose surgery may improve VA, e.g. cataract)
* Ocular treatments: treatment with anti-VEGF drugs for > 5 years in the study eye, pretreatment with brolucizumab at any time in the study eye, previous treatment with investigational drugs in the last 6 months, intraocular or periocular steroids at any time, macular laser photocoagulation or photodynamic therapy at any time, peripheral laser photocoagulation within 3 months prior to baseline, intraocular surgery within 3 months prior to baseline, vitreoretinal surgery at any time, aphakia with the absence of posterior capsule (study eye)
* Stroke or myocardial infarction during the 6 month period prior to baseline
* Systemic anti-VEGF therapy during the 3-month period prior to baseline

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (19):
- Germany (16):
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Homburg
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Neubrandenburg
  - Novartis Investigative Site, Ulm
- Switzerland (3):
  - Novartis Investigative Site, Lausanne, CHE
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Zurich

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on ww.clinicalstudydatarequest.com.
URL: http://www.clinicalstudydatarequest.com/

REFERENCES:
- [Derived] Holz FG, Schmitz-Valckenberg S, Wolf A, Agostini H, Lorenz K, Pielen A, Feltgen N, Guthoff R, Quiering C, Clemens A, Jaeger K. A randomized, open-label, multicenter study of switching to brolucizumab with or without a loading dose for patients with suboptimal anatomically controlled neovascular age-related macular degeneration-the FALCON study. Graefes Arch Clin Exp Ophthalmol. 2022 Aug;260(8):2695-2702. doi: 10.1007/s00417-022-05591-z. Epub 2022 Feb 21. PMID 35188581
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2506

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: If both eyes were eligible as per the inclusion and exclusion criteria, the eye with the worse visual acuity should have been selected for study eye, unless the investigator deemed it more appropriate to select the eye with better visual acuity, based on medical reasons or local ethical requirements.
Groups:
- Brolucizumab 6 mg Loading: 3 x 4-weekly initial injections followed by an injection every 12 weeks
Period: Overall Study
Arm/Group | Brolucizumab 6 mg Loading | Brolucizumab 6 mg Non-loading
Started | 25 | 27
Completed | 25 | 26
Not Completed | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brolucizumab 6 mg Loading | Brolucizumab 6 mg Non-loading | Total
Number analyzed (Participants) | 25 | 27 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.6 (6.3) | 77.4 (8.3) | 77.5 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 18 | 32
  Male | 11 | 9 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 25 | 27 | 52
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Week 40 to Week 52: LS Mean Change From Baseline in Best Corrected Visual Acuity (BCVA) in the Study Eye
Description: BCVA was assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts.
  Visual function of the study eye was assessed using the ETDRS protocol. Participants with a BCVA ETDRS letter score between 78 and 23 ETDRS letters (inclusive) at Screening and Baseline in the study eye were included.
  Min and max possible scores are 0-100 respectively. A higher score represents better functioning.
Time Frame: Baseline, Week 40 to Week 52
Population: full analysis set - included all patients with a valid assessment without a protocol deviation with impact
Measure: Least Squares Mean (Standard Error); unit: Letters read
Arm/Group | Brolucizumab 6 mg Loading | Brolucizumab 6 mg Non-loading
Number analyzed (Participants) | 25 | 26
Letters read
  Week 40 | 3.24 (1.32) | -0.50 (1.28)
  Week 44 | 3.88 (1.66) | -0.27 (1.60)
  Week 48 | 3.12 (1.71) | -2.23 (1.65)
  Week 52 | 2.76 (1.64) | -1.43 (1.58)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg Loading vs Brolucizumab 6 mg Non-loading; Week 40; Test type: Other — Analysis was purely descriptive; MMRM model; Difference = -3.74, 95% CI 2-sided [-7.47 to -0.01], Standard Error of Mean 1.84
Statistical Analysis 2: Comparison: Brolucizumab 6 mg Loading vs Brolucizumab 6 mg Non-loading; Week 44; Test type: Other — Analysis was purely descriptive; MMRM model; Difference = -4.15, 95% CI 2-sided [-8.78 to -0.48], Standard Error of Mean 2.30
Statistical Analysis 3: Comparison: Brolucizumab 6 mg Loading vs Brolucizumab 6 mg Non-loading; Week 48; Test type: Other — Analysis was purely descriptive; MMRM model; Difference = -5.35, 95% CI 2-sided [-10.13 to -0.58], Standard Error of Mean 2.38
Statistical Analysis 4: Comparison: Brolucizumab 6 mg Loading vs Brolucizumab 6 mg Non-loading; Week 52; Test type: Other — Analysis was purely descriptive; MMRM model; Difference = -4.19, 95% CI 2-sided [-8.77 to 0.39], Standard Error of Mean 2.28
Statistical Analysis 5: Comparison: Brolucizumab 6 mg Loading vs Brolucizumab 6 mg Non-loading; Mean of Week 40 to Week 52; Test type: Other — Analysis was purely descriptive; MMRM model; Difference = -4.36, 95% CI 2-sided [-8.56 to -0.16], Standard Error of Mean 2.09

2. Secondary Outcome: Treatment Intervals Before and During the Study
Description: Treatment interval distribution.
  Treatment interval during the study, within 24 weeks prior to baseline and interval between the last 2 injections in the study. In the loading arm, data from the loading period was excluded.
Time Frame: -24 Weeks, Baseline, Week 52
Population: full analysis set
Measure: Median (Full Range); unit: days
Arm/Group | Brolucizumab 6 mg Loading | Brolucizumab 6 mg Non-loading
Number analyzed (Participants) | 25 | 27
days
  within 24 weeks prior to baseline | 54.7 [40.0 to 152.0] | 68.5 [37.2 to 165.0]
  from baseline to week 52 (n=23,25): number analyzed (Participants) | 23 | 25
  from baseline to week 52 (n=23,25) | 64.8 [47.5 to 85.3] | 77.8 [55.8 to 85.8]
  Last treatment interval during the study (n=25,25): number analyzed (Participants) | 25 | 25
  Last treatment interval during the study (n=25,25) | 56.0 [28.0 to 88.0] | 65.0 [56.0 to 91.0]

3. Secondary Outcome: Number of Patients With Prolonged Interval
Description: Treatment interval distribution.
  Prolongation was calculated by comparing the mean treatment interval in last 24 weeks prior to first brolucizumab injection (a) with the mean of the average treatment interval during the study (loading phase excluded in the loading arm) and (b) with the last treatment interval during the study. Patients with only 1 injection during the treatment period were calculated as non-responders (no prolon-gation).
Time Frame: Baseline, Week 52
Population: full analysis set - included all patients with a valid assessment without a protocol deviation with impact
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg Loading | Brolucizumab 6 mg Non-loading
Number analyzed (Participants) | 25 | 27
Participants
  from baseline to week 52 | 18 | 12
  Last treatment interval during the study | 13 | 10

4. Secondary Outcome: Proportion of Patients Who Maintained on q12w Regimen.
Description: Treatment interval distribution up to Week 52.
  Proportion of patients maintained on q12w treatment frequency in the two brolucizumab groups up to week 52. Patients who discontinued treatment before week 52 were rated as non-responders, i.e., as patients who did not maintain the q12w regimen. In the loading arm, the loading period up to week 12 was not considered in the analysis.
Time Frame: Up to week 52
Population: full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg Loading | Brolucizumab 6 mg Non-loading
Number analyzed (Participants) | 25 | 27
Participants | 8 | 6

5. Secondary Outcome: Distribution of Patients at Every 8 Weeks / Every 12 Weeks Intervals - Frequency of Switches in Treatment Intervals Between Baseline and Week 52
Description: Treatment interval distribution
Time Frame: Up to Week 52
Population: full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg Loading | Brolucizumab 6 mg Non-loading
Number analyzed (Participants) | 25 | 27
Participants
  Switch q12w to q8w (overall) | 15 | 19
  Switch q8w to q12w (overall) | 3 | 6

6. Secondary Outcome: Mean Change in Best-corrected Visual Acuity
Description: as for outcome 1
Time Frame: Baseline, Weeks 16 to 28, Week 52
Population: full analysis set
Measure: Mean (Standard Deviation); unit: Letters read
Arm/Group | Brolucizumab 6 mg Loading | Brolucizumab 6 mg Non-loading
Number analyzed (Participants) | 25 | 27
Letters read
  Baseline | 72.0 (8.7) | 71.6 (11.5)
  Mean of weeks 16 to 28 | 74.9 (9.2) | 71.2 (12.9)
  Week 52 | 74.8 (9.1) | 69.8 (16.1)

7. Secondary Outcome: Number of Patients With Best-corrected Visual Acuity Improvements of >= 5, >= 10 and >= 15 Letters
Description: as for outcome 1
Time Frame: Baseline, up to Week 52
Population: full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg Loading | Brolucizumab 6 mg Non-loading
Number analyzed (Participants) | 25 | 27
Participants
  BCVA ≥ 5 ETDRS letters improvement during the study | 9 | 5
  BCVA ≥ 10 ETDRS letters improvement during the study | 2 | 2
  BCVA ≥ 15 ETDRS letters improvement during the study | 1 | 0

8. Secondary Outcome: Number of Patients With Best-corrected Visual Acuity >= 69 Letters
Description: as for outcome 1
Time Frame: Baseline, up to Week 52
Population: full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg Loading | Brolucizumab 6 mg Non-loading
Number analyzed (Participants) | 25 | 27
Participants | 20 | 19

9. Secondary Outcome: LS Mean Change in Best-corrected Visual Acuity From Baseline at Week 52
Description: as for outcome 1
Time Frame: Baseline, Week 52
Population: full analysis set - included all patients with a valid assessment without a protocol deviation with impact
Measure: Least Squares Mean (Standard Error); unit: Letters read
Arm/Group | Brolucizumab 6 mg Loading | Brolucizumab 6 mg Non-loading
Number analyzed (Participants) | 25 | 26
Letters read | 2.76 (1.64) | -1.43 (1.58)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg Loading vs Brolucizumab 6 mg Non-loading; Week 52; Test type: Other — Analysis was purely descriptive; MMRM model; Difference = -4.19, 95% CI 2-sided [-8.77 to -0.39], Standard Error of Mean 2.28

10. Secondary Outcome: Change in Central Subfield Thickness From Baseline at Weeks 12, 16, 28 and 52
Description: Change in central subfield thickness was measured by Spectral domain optical coherence tomography.
Time Frame: Baseline, Weeks 12, 16, 28 and 52
Population: full analysis set
Measure: Median (Full Range); unit: µm
Arm/Group | Brolucizumab 6 mg Loading | Brolucizumab 6 mg Non-loading
Number analyzed (Participants) | 25 | 27
µm
  Week 12 | -74.0 [-275 to 27] | -8.5 [-232 to 650]
  Week 16 | -20.0 [-240 to 208] | -51.0 [-317 to 80]
  Week 28 | -21.0 [-273 to 393] | -53.0 [-357 to 60]
  Week 52 | -15.0 [-268 to 269] | -49.5 [-359 to 30]

11. Secondary Outcome: Absence of Intraretinal Fluid in the Central Subfield
Description: Change in fluids was measured by Spectral domain optical coherence tomography.
Time Frame: Every 4 weeks from baseline up to Week 52
Population: full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg Loading | Brolucizumab 6 mg Non-loading
Number analyzed (Participants) | 25 | 27
Participants
  Baseline | 13 | 16
  Week 4 | 19 | 22
  Week 8 | 17 | 16
  Week 12 | 21 | 16
  Week 16 | 12 | 21
  Week 20 | 16 | 20
  Week 24 | 17 | 18
  Week 28 | 16 | 20
  Week 32 | 18 | 17
  Week 36 | 17 | 17
  Week 40 | 16 | 21
  Week 44 | 16 | 19
  Week 48 | 19 | 19
  Week 52 | 16 | 21

12. Secondary Outcome: Absence of Subretinal Fluid in the Central Subfield
Description: Change in fluids was measured by Spectral domain optical coherence tomography.
Time Frame: Every 4 weeks from baseline up to Week 52
Population: full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg Loading | Brolucizumab 6 mg Non-loading
Number analyzed (Participants) | 25 | 27
Participants
  Baseline | 5 | 6
  Week 4 | 13 | 18
  Week 8 | 18 | 12
  Week 12 | 20 | 6
  Week 16 | 8 | 15
  Week 20 | 3 | 12
  Week 24 | 13 | 12
  Week 28 | 9 | 13
  Week 32 | 11 | 14
  Week 36 | 11 | 14
  Week 40 | 10 | 15
  Week 44 | 8 | 10
  Week 48 | 10 | 15
  Week 52 | 9 | 16

13. Secondary Outcome: Absence of Sub-retinal Pigment Epithelium Fluid in the Central Subfield
Description: Change in fluids was measured by Spectral domain optical coherence tomography.
Time Frame: Every 4 weeks from baseline up to Week 52
Population: full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg Loading | Brolucizumab 6 mg Non-loading
Number analyzed (Participants) | 25 | 27
Participants
  Baseline | 15 | 13
  Week 4 | 20 | 21
  Week 8 | 18 | 16
  Week 12 | 20 | 17
  Week 16 | 20 | 14
  Week 20 | 17 | 16
  Week 24 | 18 | 16
  Week 28 | 19 | 21
  Week 32 | 19 | 20
  Week 36 | 18 | 19
  Week 40 | 22 | 18
  Week 44 | 18 | 18
  Week 48 | 21 | 18
  Week 52 | 17 | 16

14. Secondary Outcome: Presence of Active Choroidal Neovascularization Leakage
Description: Presence of active choroidal neovascularization leakage was measured by Fluorescein angiography.
  CNV = choroidal neovascularization; MNV = macular neovascularization
Time Frame: At Week 52
Population: full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg Loading | Brolucizumab 6 mg Non-loading
Number analyzed (Participants) | 25 | 27
Participants
  Active CNV leakage at week 52 - Yes | 17 | 15
  Active CNV leakage at week 52 - No | 7 | 10
  Active CNV leakage at week 52 - missing | 1 | 2
  CNV location at week 52 - Subfoveal | 11 | 10
  CNV location at week 52 - Extrafoveal | 6 | 5
  CNV location at week 52 - Not applicable | 7 | 10
  CNV location at week 52 - Missing | 1 | 2
  CNV subtype at week 52 - Type 1 MNV | 12 | 9
  CNV subtype at week 52 - Mixed type 1 and type 2 MNV | 2 | 1
  CNV subtype at week 52 -Type 3 MNV | 3 | 5
  CNV subtype at week 52 - Not applicable | 7 | 10
  CNV subtype at week 52 - Missing | 1 | 2

15. Secondary Outcome: Overview of TEAEs
Description: An adverse event (AE) is any untoward medical occurrence (e.g. any unfavorable and unintended sign (including abnormal laboratory findings), symptom or disease) in a subject or clinical investigation subject after providing written informed consent for participation in the study.
  Treatment-emergent AEs are AEs that developed on or after first study treatment administration, or any event previously present that worsened following exposure to the study treatment.
Time Frame: Adverse events are reported from first dose of study treatment until end of study treatment plus 30 days post treatment, up to a maximum timeframe of approximately 52 weeks.
Population: safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg Loading | Brolucizumab 6 mg Non-loading
Number analyzed (Participants) | 25 | 27
Participants
  Any AE | 23 | 26
  Ocular AE(s) in the study eye | 17 | 19
  Ocular AE(s) in the fellow eye | 4 | 9
  Non-ocular AE(s) | 20 | 19
  AE(s) related to injection procedure | 11 | 12
  AE(s) related to study drug | 9 | 12
  SAE(s) | 5 | 6
  Ocular SAE(s) in the study eye | 1 | 4
  Non-ocular SAE(s) | 4 | 2
  Death | 0 | 1
  Non-fatal SAE(s) | 5 | 6
  Discontinuation of study treatment due to any AE(s) | 2 | 5
  Discontinuation of study treatment due to non-serious AE(s) | 0 | 4
  Discontinuation of study treatment due to any SAE(s) | 2 | 2

16. Secondary Outcome: Ocular TEAEs in the Study Eye by Primary System Organ Class
Description: as for outcome 15
Time Frame: as for outcome 15
Population: safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg Loading | Brolucizumab 6 mg Non-loading
Number analyzed (Participants) | 25 | 27
Participants
  Total | 17 | 19
  Eye disorders | 16 | 17
  General disorders and administration site conditions | 0 | 1
  Infections and infestations | 2 | 2
  Injury, poisoning and procedural complications | 2 | 1
  Investigations | 2 | 4

17. Secondary Outcome: Ocular TEAEs in the Study Eye by Preferred Term (at Least 5% in Any Group)
Description: as for outcome 15
Time Frame: as for outcome 15
Population: safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg Loading | Brolucizumab 6 mg Non-loading
Number analyzed (Participants) | 25 | 27
Participants
  Conjunctival haemorrhage | 7 | 5
  Visual acuity reduced | 2 | 3
  Eye inflammation | 1 | 3
  Intraocular pressure increased | 1 | 3
  Retinal oedema | 1 | 3
  Dry Eye | 1 | 2
  Neovascular age-related macular degeneration | 1 | 2
  Vitreous detachment | 2 | 1
  Cataract | 0 | 2
  Conjunctivitis | 0 | 2
  Retinal exudates | 0 | 2
  Vitreous floaters | 0 | 2

18. Secondary Outcome: Non-ocular TEAEs - Total
Description: as for outcome 15
Time Frame: as for outcome 15
Population: safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg Loading | Brolucizumab 6 mg Non-loading
Number analyzed (Participants) | 25 | 27
Participants | 20 | 19

19. Secondary Outcome: Ocular TEAEs in the Study Eye of Moderate or Severe Intensity
Description: as for outcome 15
Time Frame: as for outcome 15
Population: safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg Loading | Brolucizumab 6 mg Non-loading
Number analyzed (Participants) | 25 | 27
Participants
  Any AE of moderate intensity | 3 | 8
  Cataract - moderate intensity | 0 | 2
  Conjunctival haemorrhage - moderate intensity | 0 | 1
  Conjunctival irritation - moderate intensity | 1 | 0
  Conjunctivitis allergic - moderate intensity | 0 | 1
  Dry eye - moderate intensity | 1 | 1
  Eye inflammation - moderate intensity | 0 | 1
  Eye pain - moderate intensity | 0 | 1
  Neovascular age-related macular degeneration - moderate intensity | 0 | 1
  Retinal vasculitis - moderate intensity | 0 | 2
  Subretinal fluid - moderate intensity | 0 | 1
  Visual acuity reduced - moderate intensity | 1 | 0
  Vital dye staining cornea present - moderate intensity | 0 | 1
  Vitreous opacities - moderate intensity | 0 | 1
  Any AE of severe intensity | 1 | 2
  Endophthalmitis - severe intensity | 1 | 0
  Eye inflammation - severe intensity | 1 | 1
  Intraocular pressure increased - severe intensity | 0 | 1
  Retinal haemorrhage - severe intensity | 0 | 1
  Retinal neovascularization - severe intensity | 0 | 1
  Visual acuity reduced - severe intensity | 0 | 1

20. Post Hoc Outcome: All Collected Deaths
Description: On-treatment deaths are reported from first dose of study treatment until end of study treatment plus 30 days after last treatment, up to a maximum timeframe of approximately 52 weeks.
  Post-treatment death data are reported from day 31 after last treatment to end of study (Week 52).
Time Frame: Fatality data are reported from first dose of study treatment until approximately Week 52.
Population: safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg Loading | Brolucizumab 6 mg Non-loading
Number analyzed (Participants) | 25 | 27
Participants
  On-treatment Deaths | 0 | 0
  Post-treatment Deaths | 0 | 1
  Total Deaths | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse events are reported from first dose of study treatment until end of study treatment plus 30 days post treatment, up to a maximum timeframe of approximately 52 weeks.
Arm/Group | Brolucizumab 6 mg Loading | Brolucizumab 6 mg Non-loading
All-Cause Mortality (participants affected / at risk) | 0/25 | 1/27
Serious Adverse Events (participants affected / at risk) | 5/25 | 6/27
Other Adverse Events (participants affected / at risk) | 23/25 | 26/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brolucizumab 6 mg Loading (N=25) | Brolucizumab 6 mg Non-loading (N=27)
Eye inflammation- Study Eye (Eye disorders) | 1 | 1
Iridocyclitis- Study Eye (Eye disorders) | 0 | 1
Retinal haemorrhage- Study Eye (Eye disorders) | 0 | 1
Retinal neovascularisation- Study Eye (Eye disorders) | 0 | 1
Retinal vasculitis- Study Eye (Eye disorders) | 0 | 1
Visual acuity reduced- Study Eye (Eye disorders) | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Endophthalmitis- Study Eye (Infections and infestations) | 1 | 0
Kidney infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Intraocular pressure increased- Study Eye (Investigations) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Chromophobe renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ballismus (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brolucizumab 6 mg Loading (N=25) | Brolucizumab 6 mg Non-loading (N=27)
Anterior chamber cell- Study Eye (Eye disorders) | 1 | 0
Blepharitis- Bilateral (Eye disorders) | 0 | 1
Cataract- Bilateral (Eye disorders) | 0 | 1
Cataract- Study Eye (Eye disorders) | 0 | 1
Chalazion- Study Eye (Eye disorders) | 1 | 0
Conjunctival haemorrhage- Study Eye (Eye disorders) | 7 | 5
Conjunctival hyperaemia- Fellow Eye (Eye disorders) | 0 | 1
Conjunctival irritation- Study Eye (Eye disorders) | 1 | 0
Conjunctivitis allergic- Bilateral (Eye disorders) | 0 | 2
Corneal epithelial microcysts- Study Eye (Eye disorders) | 0 | 1
Corneal erosion- Study Eye (Eye disorders) | 1 | 0
Detachment of retinal pigment epithelium- Study Eye (Eye disorders) | 0 | 1
Dry eye- Bilateral (Eye disorders) | 1 | 2
Eczema eyelids- Fellow Eye (Eye disorders) | 0 | 1
Eczema eyelids- Study Eye (Eye disorders) | 0 | 1
Episcleritis- Study Eye (Eye disorders) | 0 | 1
Eye inflammation- Bilateral (Eye disorders) | 0 | 1
Eye inflammation- Study Eye (Eye disorders) | 0 | 2
Eye irritation- Study Eye (Eye disorders) | 1 | 0
Eye pain (Eye disorders) | 0 | 1
Eye pain- Study Eye (Eye disorders) | 0 | 1
Eye ulcer- Fellow Eye (Eye disorders) | 0 | 1
Foreign body sensation in eyes- Study Eye (Eye disorders) | 0 | 1
Macular oedema- Fellow Eye (Eye disorders) | 0 | 1
Macular oedema- Study Eye (Eye disorders) | 1 | 1
Neovascular age-related macular degeneration- Fellow Eye (Eye disorders) | 3 | 1
Neovascular age-related macular degeneration- Study Eye (Eye disorders) | 1 | 2
Ocular hyperaemia- Fellow Eye (Eye disorders) | 1 | 0
Posterior capsule opacification- Fellow Eye (Eye disorders) | 0 | 1
Retinal aneurysm- Fellow Eye (Eye disorders) | 0 | 1
Retinal aneurysm- Study Eye (Eye disorders) | 0 | 1
Retinal cyst- Fellow Eye (Eye disorders) | 0 | 2
Retinal exudates- Bilateral (Eye disorders) | 0 | 1
Retinal exudates- Study Eye (Eye disorders) | 0 | 1
Retinal haemorrhage- Study Eye (Eye disorders) | 1 | 1
Retinal oedema- Fellow Eye (Eye disorders) | 0 | 1
Retinal oedema- Study Eye (Eye disorders) | 1 | 3
Retinal vasculitis- Study Eye (Eye disorders) | 0 | 2
Retinopathy hypertensive (Eye disorders) | 1 | 0
Scleritis- Study Eye (Eye disorders) | 0 | 1
Subretinal fibrosis- Study Eye (Eye disorders) | 0 | 1
Subretinal fluid- Fellow Eye (Eye disorders) | 1 | 1
Subretinal fluid- Study Eye (Eye disorders) | 1 | 1
Vision blurred- Study Eye (Eye disorders) | 0 | 1
Visual acuity reduced- Bilateral (Eye disorders) | 1 | 0
Visual acuity reduced- Fellow Eye (Eye disorders) | 0 | 1
Visual acuity reduced- Study Eye (Eye disorders) | 1 | 3
Vitreal cells- Study Eye (Eye disorders) | 0 | 1
Vitreous detachment- Study Eye (Eye disorders) | 2 | 1
Vitreous floaters- Bilateral (Eye disorders) | 0 | 1
Vitreous floaters- Study Eye (Eye disorders) | 0 | 2
Vitreous haemorrhage- Fellow Eye (Eye disorders) | 1 | 0
Vitreous opacities- Study Eye (Eye disorders) | 0 | 1
Tooth impacted (Gastrointestinal disorders) | 0 | 1
Application site wound (General disorders) | 0 | 1
Injection site pain- Study Eye (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 1
Retention cyst- Fellow Eye (General disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1
COVID-19 (Infections and infestations) | 6 | 5
Conjunctivitis- Study Eye (Infections and infestations) | 0 | 2
Cystitis (Infections and infestations) | 1 | 2
Gastrointestinal viral infection (Infections and infestations) | 1 | 0
Herpes virus infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Hordeolum- Study Eye (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Lyme disease (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 6 | 5
Oral herpes (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Sialoadenitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0
Bone contusion (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 1 | 0
Expired product administered- Study Eye (Injury, poisoning and procedural complications) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 2
Intra-ocular injection complication- Fellow Eye (Injury, poisoning and procedural complications) | 0 | 1
Intra-ocular injection complication- Study Eye (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Stress fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood pressure increased (Investigations) | 2 | 0
Intraocular pressure increased- Fellow Eye (Investigations) | 0 | 1
Intraocular pressure increased- Study Eye (Investigations) | 1 | 2
Vital dye staining cornea present- Study Eye (Investigations) | 1 | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Jaw cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Blepharal papilloma- Fellow Eye (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Incontinence (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Palmar erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 3 | 3
Hypertensive crisis (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-11-30): https://cdn.clinicaltrials.gov/large-docs/35/NCT04679935/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-25): https://cdn.clinicaltrials.gov/large-docs/35/NCT04679935/SAP_001.pdf